CLINICAL TRIAL: NCT01277627
Title: Influence of Nevirapine on HCV Viral Load Among HIV/HCV-coinfected Patients
Brief Title: Influence of Nevirapine on HCV Viral Load
Acronym: HELICON
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Valme University Hospital (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: JOSE ANTONIO MIRA-ESCARTI, INFECTIOUS DISEASES UNIT, VALME UNIVERSITY HOSPITAL, SEVILLE, SPAIN
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: JAP-NEV-2010-01
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2010-12

CONDITIONS: HCV Infection.; HCV Viral Load.
Keywords: HCV; HIV; Nevirapine; HCV viral load; Efavirenz; Protease inhibitors
MeSH Terms: conditions — Hepatitis C | interventions — Nevirapine; efavirenz; Protease Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nevirapine (Active Comparator)
  Interventions: Drug: Nevirapine; Drug: efavirenz, protease inhibitors
- Non-nevirapine (Active Comparator)
  Interventions: Drug: Nevirapine; Drug: efavirenz, protease inhibitors

INTERVENTIONS:
Drug: Nevirapine — nevirapine: 400 mg a day.
Drug: efavirenz, protease inhibitors — efavirenz: 600 mg a day

SUMMARY:
Nevirapine-based antiretroviral therapy is associated with lower plasma HCV viral load in HIV/HCV-coinfected individuals.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection.
* Older than 18 years.
* Chronic hepatitis C.
* Undetectable HIV viral load during one year before starting study.
* To have not received HCV therapy during one year before starting study.
* To have not started efavirenz or protease inhibitors o nucleoside analogs during 6 months before starting study.
* Non contraindications for drugs included in this study.
* To change an antiretroviral regimen including efavirenz or protease inhibitors by nevirapine due to side effects, interactions or pregnancy (NVP group)
* To continue with a antiretroviral regimen including efavirenz or protease inhibitors (non-NVP group)

Both groups will be matched according to these variables:

* Liver stiffness.
* HCV genotype.
* Hospital.
* Time from starting antiretroviral therapy.
* Previous third drug (EFV or PI) to introduction of NVP.

Exclusion Criteria:

* HCV therapy during follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Changes in HCV viral load | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Valme University Hospital, Seville, Seville, Spain